CLINICAL TRIAL: NCT04670744
Title: Retrospective Analysis for the Identification of Outcome Relevant Indicators ("Patterns") in Routine Data and Investigation of the Influence on Patient-centered Outcome for a Data-driven Improvement of Quality-based Treatment of Perioperative and Intensive Care Patients
Brief Title: Identification of Outcome Relevant Indicators in Routine Data
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: QUALIPATT
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Anesthesiological Risk Reduction; Intensive Care Risk Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The availability of electronic documentation systems in patient care means that large amounts of clinical routine data are available from which conclusions can be drawn for improving patient care. Compared to conventional research approaches, a data science-oriented approach offers the possibility of identifying patterns in routine data ("pattern recognition") that are relevant for patient-centered outcomes.

Numerous projects and sub-projects can be evaluated from this data set.

DETAILED DESCRIPTION:
The patterns that are relevant for patient-centered outcomes can be combinations of different parameters (e.g. vital signs, laboratory values, previous illnesses), which in themselves do not necessarily have a pathogenic effect, but in a specific combination may have a high relevance for the patient-centered outcome.

This project pursues as research goal the anesthesiological and intensive care risk reduction. To this end, the existing data sets of routine care are to be used to identify outcome-relevant patterns in order to derive recommendations for improving treatment in line with the patient's wishes. Standard Operating Procedures (SOPs) and Quality Indicators (QIs) in combination with the data of routine clinical care will be used as a basis. The approach outlined is closely linked to the development of quality-based treatment structures. In order to be able to offer medical treatment at a high level, associated processes must be known and operationalized, i.e. measurable. QIs (quality indicators) are an established instrument for measuring individual dimensions of treatment quality, and our clinic is a leading participant in this process at both national and international level (see Spies et al. Guidelines for Delirium, Analgesia and Sedation). The mapping of quality-based treatment structures as SOPs (Standard Operating Procedures) is also essential in this context (see Spies et al. SOPs in Anesthesiology and Pain Therapy, Thieme Verlag). By applying data science-based methods, this study pursues the overall goal of supporting the transfer of evidence-based findings in the form of QIs and SOPs into patient care.

Numerous projects and sub-projects can be evaluated from this data set.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0 to 120 years
* Gender: female, male, diverse
* Electronically documented anesthesiological or intensive care treatment in the HIS (Hospital Information System) and PDMS (Patient Data Management System) of the Charité (Department of Anesthesiology and Intensive Care Medicine, CCM/CVK/CBF) since 2016

Exclusion Criteria:

-none

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: At the department for anesthesiology with a focus on operative intensive care medicine, approximately 60,000 anaesthesias are performed annually. The data sets of documentation systems used in this context date back approximately to the year 2016 and are to be considered for the development of data science-based models depending on selected QI or SOPs.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional status | 01.01.2016-31.12.2024
  The functional status of the patient is measured by routine score data. The scores, which measure physical, role, and social functioning, and mobility reflect worse/better outcome depending on the score construction.

SECONDARY OUTCOMES:
Morbidity | 01.01.2016-31.12.2024
  Morbidity is evaluated by International Classification of Diseases (ICD) (10th version). /Operation codes (OPS)
Mortality I | 01.01.2016-31.12.2024
  Mortality is measured by inhouse mortality
Mortality II | 01.01.2016-31.12.2025
  Mortality is measured by long-term mortality (1 year)
Accounting data | 01.01.2016-31.12.2024
  Accounting data are providid by the controlling department

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No